CLINICAL TRIAL: NCT02759471
Title: One Month Dispensing Study Comparing the Clinical Performance of the Comfilcon A Sphere Lenses Compared to Comfilcon A Asphere Lenses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: EX-MKTG-63
Record Dates: First submitted 2016-04-29; First posted 2016-05-03 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- comfilcon A asphere (test) (Experimental): Habitual wearers of comfilcon A sphere lens (control) are refitted with comfilcon A asphere lens (test).
  Interventions: Device: comfilcon A asphere lens (test)
- comfilcon A sphere (control) (Active Comparator): Habitual wearers of comfilcon A sphere lens (control) are refitted with comfilcon A asphere lens (test).
  Interventions: Device: comfilcon A sphere lens (control)

INTERVENTIONS:
Device: comfilcon A sphere lens (control) — contact lens
  Arms: comfilcon A sphere (control)
Device: comfilcon A asphere lens (test) — contact lens
  Arms: comfilcon A asphere (test)

SUMMARY:
This is a prospective, multi-center, subject-masked, bilateral wear, one month dispensing study comparing the clinical performance of the subjects' habitual comfilcon A sphere lens (control) following a refit with comfilcon A asphere lens (test). After the dispensing visit, subjects will return for follow-up evaluations after 2 weeks, and 1 month.

DETAILED DESCRIPTION:
This is a prospective, multi-center, subject-masked, bilateral wear, one month dispensing study comparing the clinical performance of the subjects' habitual comfilcon A sphere lens (control) following a refit with comfilcon A asphere lens (test). After the dispensing visit, subjects will return for follow-up evaluations after 2 weeks, and 1 month.

Both comfilcon A sphere lens (control) and comfilcon A asphere lens (test) are Coopervison lenses.

ELIGIBILITY:
Inclusion criteria

A person is eligible for inclusion in the study if he/she:

* Is between 18 and 34 years of age (inclusive)
* Has had a self-reported eye exam in the last two years
* Is an adapted comfilcon A sphere contact lens wearer
* Uses digital devices, (e.g. computer, tablet, smart phone, iPad), for more than 4 hours a day, 5 days a week.
* Has a contact lens spherical prescription between -1.00 to -6.00 (inclusive)
* Has a spectacle cylinder no greater than 0.75D (Diopters) in each eye.
* Can achieve best corrected spectacle distance visual acuity of 20/25 (0.10 logMAR) or better in each eye.
* Can achieve a distance visual acuity of 20/30 (0.18 logMAR) or better in each eye with the study contact lenses.
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter.
* Has a contact lens refraction that fits within the available parameters of the study lenses.
* Is willing to comply with the wear schedule (at least 5 days per week, > 8 hours/day assuming there are no contraindications for doing so).
* Is willing to comply with the visit schedule

Exclusion Criteria

A person will be excluded from the study if he/she:

* Has a history of not achieving comfortable CL (Contact Lens) wear (5 days per week; > 8 hours/day)
* Presents with clinically significant anterior segment abnormalities
* Presents with ocular or systemic disease or need of medications which might interfere with contact lens wear.
* Presents with slit lamp findings that would contraindicate contact lens wear such as:

  * Pathological dry eye or associated findings
  * Significant pterygium, pinguecula, or corneal scars within the visual axis
  * Neovascularization > 0.75 mm in from of the limbus
  * Giant papillary conjunctivitis (GCP) worse than grade 1
  * Anterior uveitis or iritis (or history in past year)
  * Seborrheic eczema of eyelid region, Seborrheic conjunctivitis
  * History of corneal ulcers or fungal infections
  * Poor personal hygiene
* Has a known history of corneal hypoesthesia (reduced corneal sensitivity)
* Has aphakia, keratoconus or a highly irregular cornea.
* Has presbyopia or has dependence on spectacles for near work over the contact lenses.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.
* Is habitually using rewetting/ lubricating eye drops (more than once per day)

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Sacco, OD, Principal Investigator — Sacco Eye Group; Gina Wesley, OD, Principal Investigator — Complete Eye Care of Medina; Thomas Quinn, OD, MS, FAAO, Principal Investigator — Drs. Quinn, Foster, & Associates; David Ardaya, OD, Principal Investigator — Golden Optometric Group
Locations (4):
- United States (4):
  - Golden Optometric Group, Whittier, California
  - Complete Eye Care of Medina, Medina, Minnesota
  - Sacco Eye Group, Vestal, New York
  - Drs. Quinn, Foster, & Associates, Athens, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Comfilcon A Sphere (Control) and Comfilcon A Asphere (Test): Habitual wearers of comfilcon A sphere lens (control) are refitted with comfilcon A asphere lens (test).
  comfilcon A sphere lens (control): contact lens
  comfilcon A asphere lens (test): contact lens
Period: Overall Study
Arm/Group | Comfilcon A Sphere (Control) and Comfilcon A Asphere (Test)
Started | 54
Completed | 52
Not Completed | 2
Not completed — discomfort | 2

BASELINE CHARACTERISTICS:
Arm/Group | Comfilcon A Sphere (Control) and Comfilcon A Asphere (Test)
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] | 26 [18 to 34]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Lens Fit - Centration
Description: Lens fit evaluation of centration for comfilcon A sphere and comfilcon A asphere lens. (Scale: optimum, decentration acceptable and decentration unacceptable).
Time Frame: baseline, 2 weeks, 1 month
Population: One participants data for both the 2 week and 1 month visit was not included due to participant protocol deviation.
Measure: Number; unit: participants
Groups:
- Comfilcon A Sphere (Control); Comfilcon A Asphere (Test): habitual wearers of comfilcon A sphere are refitted with comfilcon A asphere
Arm/Group | Comfilcon A Sphere (Control) | Comfilcon A Asphere (Test)
Number analyzed (Participants) | 52 | 52
participants
  Baseline, Optimum | 48 | 46
  Baseline, Acceptable | 4 | 6
  Baseline, Unacceptable | 0 | 0
  At 2 weeks, optimum: number analyzed (Participants) | 51 | 51
  At 2 weeks, optimum | NA — participants were refitted with test lens and habitual lens were not evaluated at this time point. | 45
  At 2 weeks, acceptable: number analyzed (Participants) | 51 | 51
  At 2 weeks, acceptable | NA — participants were refitted with test lens and habitual lens were not evaluated at this time point. | 6
  At 2 weeks, unacceptable: number analyzed (Participants) | 51 | 51
  At 2 weeks, unacceptable | NA — participants were refitted with test lens and habitual lens were not evaluated at this time point. | 0
  At 1 month, optimum: number analyzed (Participants) | 51 | 51
  At 1 month, optimum | NA — participants were refitted with test lens and habitual lens were not evaluated at this time point. | 46
  At 1 month, acceptable: number analyzed (Participants) | 51 | 51
  At 1 month, acceptable | NA — participants were refitted with test lens and habitual lens were not evaluated at this time point. | 5
  At 1 month, unacceptable: number analyzed (Participants) | 51 | 51
  At 1 month, unacceptable | NA — participants were refitted with test lens and habitual lens were not evaluated at this time point. | 0

2. Primary Outcome: Lens Fit - Corneal Coverage
Description: Lens fit evaluation of corneal coverage for comfilcon A sphere and comfilcon A asphere lens. ('yes' - full coverage, or 'no' - incomplete corneal coverage).
Time Frame: baseline, 2 weeks, 1 month
Population: One participants data for both the 2 week and 1 month visit was not included due to participant protocol deviation.
Measure: Number; unit: participants
Arm/Group | Comfilcon A Sphere (Control) | Comfilcon A Asphere (Test)
Number analyzed (Participants) | 52 | 52
participants
  Baseline, yes | 52 | 52
  2 weeks, yes: number analyzed (Participants) | 51 | 51
  2 weeks, yes | 51 | 51
  1 month, yes: number analyzed (Participants) | 51 | 51
  1 month, yes | 51 | 51

3. Primary Outcome: Lens Fit - Post-blink Movement
Description: Lens fit evaluation of post-blink movement for comfilcon A sphere and comfilcon A asphere lens. (Scale 0-4, 0=Insufficient, unacceptable movement, 1=Minimal, but acceptable movement, 2=Optimal movement, 3=Moderate, but acceptable movement, 4=Excessive, unacceptable movement).
Time Frame: baseline, 2 weeks, 1 month
Population: One participants data for both the 2 week and 1 month visit was not included due to participant protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A Sphere (Control) | Comfilcon A Asphere (Test)
Number analyzed (Participants) | 52 | 52
units on a scale
  Baseline | 1.9 (0.6) | 1.9 (0.3)
  After 2 weeks: number analyzed (Participants) | 51 | 51
  After 2 weeks | NA (NA) — participants were refitted with test lens and habitual lens were not evaluated at this time point. | 1.9 (0.4)
  After 1 month: number analyzed (Participants) | 51 | 51
  After 1 month | NA (NA) — participants were refitted with test lens and habitual lens were not evaluated at this time point. | 1.9 (0.5)

4. Primary Outcome: Lens Preference/Acceptability
Description: Investigators preference/acceptability for comfilcon A sphere and comfilcon A asphere lenses. (Choices: strongly prefer study lenses, slightly prefer study lenses, slightly prefer habitual lenses, strongly prefer habitual lenses).
Time Frame: baseline, 2 weeks, 1 month
Measure: Number; unit: participants
Groups:
- Investigator Rating of Fit Preference: habitual wearers of comfilcon A sphere are refitted with comfilcon A asphere
Arm/Group | Investigator Rating of Fit Preference
Number analyzed (Participants) | 52
participants
  Strongly prefer comfilcon A asphere | 5
  Slightly prefer comfilcon A asphere | 39
  Strongly prefer comfilcon A sphere | 8
  Slightly prefer comfilcon A sphere | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Comfilcon A Sphere (Control) and Comfilcon A Asphere (Test)
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and the Sponsor that restricts the PI's rights to discuss or publish trial results after the trial is completed.